CLINICAL TRIAL: NCT03141944
Title: Improvement of Hypodopaminergic Syndrome With Dopaminergic Treatment in Early Parkinson's Disease
Brief Title: Evolution of Hypodopaminergic Syndrome in Early Parkinson's Disease
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.184
Record Dates: First submitted 2017-03-29; First posted 2017-05-05 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease; Apathy
Keywords: non motor symptoms
MeSH Terms: conditions — Parkinson Disease; Lethargy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apathetic patients: De novo Parkinson's Disease patients with Apathy which participated in a former study and are under dopaminergic treatment at inclusion.
  All patients will be evaluated with regard to apathy, depression, pain, behavior and personality. Primary outcome measure is the degree of Apathy by the "Starkstein scale of apathy"
  Interventions: Other: Starkstein scale of Apathy
- Non-apathetic patients: De novo Parkinson's Disease patients without Apathy which participated in a former study and are under dopaminergic treatment at inclusion.
  All patients will be evaluated with regard to apathy, depression, pain, behavior and personality. Primary outcome measure is the degree of Apathy by the "Starkstein scale of apathy"
  Interventions: Other: Starkstein scale of Apathy

INTERVENTIONS:
Other: Starkstein scale of Apathy — The degree of apathy will be evaluated with the "Starkstein scale of Apathy"

SUMMARY:
The objective of this study is to describe the evolution of hypodopaminergic syndrome in patients with Parkinson's disease.

DETAILED DESCRIPTION:
All patients to be included have been clinically described in the early phase of their disease, before instauration of dopaminergic treatment, in the context of a former study ("Non Motor Aspects in De Novo Parkinson's Disease (Honeymoon) NCT02786667") between june 2012 and june 2016.

3 to 5 years after this study, those patients who started dopaminergic treatment will be evaluated again.

The objective of this study, which takes place 3 to 5 year after the initial evaluation, is to measure the evolution of apathy and other symptoms of the hypodopaminergic syndrome.

Secondary objectives are the evolution of other parameters including pain, personality and behavior. All parameters measured have been determined of each patient in the Honeymoon study.

ELIGIBILITY:
Inclusion Criteria:

* patients who participated in "Non Motors Aspects in De Novo Parkinson's Disease (Honeymoon)" NCT02786667
* Patients under dopaminergic treatment, with stable dopaminergic treatment for at least 2 months
* Patients with medical insurance
* signed informed consent

Exclusion Criteria:

* diagnosis other than Parkinson's Disease
* dementia (Mattis <130)
* patients protected by law (i.e. pregnant or parturient women)

Ages: 33 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinon's disease who participated in "Non Motors Aspects in De Novo Parkinson's Disease (Honeymoon)" NCT02786667 between june 2012 and june 2016
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Evolution of apathy in Parkinson's disease | 1day
  Evolution of apathy in Patients with Parkinson's disease under dopaminergic treatment. The degree of apathy is evaluated with the "Starkstein Scale of Apathy".

SECONDARY OUTCOMES:
Evolution of hypodopaminergia in Parkinson's disease | 1 day
  Evolution of hypodopaminergic symptoms in Patients with Parkinson's disease under dopaminergic treatment. Hypodopaminergic symptoms are evaluated with different scales: ECMP (behavioral evaluation in Parkinsons's disease) for depression and anxiety, STAI (State-trait-anxiety inventory, self-assessment-questionnaire for anxiety, BDI (Beck depression inventory) for depression, PFS-16 (Piper Fatigue Sale) for fatigue. Hypodopaminergia is the expressed as the sum of its symptoms.
Apparition of hyperdopaminergic symptoms in Parkinson's disease | 1 day
  Apparition of hyperdopaminergic symptoms in patients with Parkinson's disease under dopaminergic treatment, with the questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP) and the ECMP scale.
Evolution of impulsivity in Parkinson's disease | 1 day
  Evolution of impulsivity in patients with Parkinson's disease under dopaminergic treatment. Evaluation with a self-assessment-questionnaire (UPPS Impulsive Behavior Scale)
Evolution of personality in Parkinson's disease | 1 day
  Evolution of personality in patients with Parkinson's disease under dopaminergic treatment with the self-assesment-questionnaire "Temperament and Character Inventory" (TCI).
Evolution of pain in Parkinson's disease | 1 day
  Evolution of pain in patients with Parkinson's disease under dopaminergic treatment with the self-assessment-questionnaire NPSI (Neuropathic Pain Symptom Inventory).
Evolution of quality of life in Parkinson's disease | 1 day
  Evolution of quality of life in patients with Parkinson's disease under dopaminergic treatment with the self-assessment-questionnaire PDQ39 (Parkinson's disease questionnaire).
Evolution of somnolence in Parkinson's disease | 1 day
  Evolution of somnolence in patients with Parkinson's disease under dopaminergic treatment with the ECMP scale.
Evolution of eating behavior in Parkinson's disease | 1 day
  Evolution of eating behavior in patients with Parkinson's disease under dopaminergic treatment with the self-assesment-questionnaire "Dutch Eating Behavior Questionnaire" - DEBQ.

CONTACTS AND LOCATIONS:
Overall Officials: Anna CASTRIOTO, MD, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - University Hospital of Grenoble, Grenoble
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - Centre Expert Régional pour la maladie de Parkinson, Poitiers
  - Hôpital de Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No